CLINICAL TRIAL: NCT00092469
Title: A Registration Study of the Safety, Tolerability, and Immunogenicity of V441 in Healthy Infants in Taiwan
Brief Title: Study of an Investigational Vaccine in Healthy Infants in Taiwan (V441-001)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V441-001; 2004_079
Record Dates: First submitted 2004-09-22; First posted 2004-09-27 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Diphtheria; Tetanus; Pertussis; Hepatitis B; Poliomyelitis
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Poliomyelitis | interventions — Tetanus Toxoid; Hepatitis B Vaccines

INTERVENTIONS:
Biological: V441, diptheria, tetanus, acellular pertussis, inactivated poliomyelitis, hepatitis B (recombinant), & Haemophilus influenza type b conjugate vaccine
  Other Names: V441

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and immune response of an investigational vaccine being evaluated to reduce the incidence of diphtheria, pertussis, tetanus, hepatitis B, poliomyelitis, and Haemophilus influenza type b.

DETAILED DESCRIPTION:
The duration of treatment is 65 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infant who received Hepatitis B vaccine within 5 days of birth and whose mother is negative to Hepatitis B surface antigen

Exclusion Criteria:

* Problems with immune system
* Recent illness with fever

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 151
Dates: Start 2002-03; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Tolerability and immune responses adequate to be protective against diphtheria, tetanus, pertussis, polio, Haemophilus Influenzae Type B, and Hepatitis B.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC